CLINICAL TRIAL: NCT05097417
Title: A Prospective Open-Label Randomized Study of Traditional Chinese Medicine Combined With Thermal and Cold Ablation for Early-stage Lung Cancer
Brief Title: Traditional Chinese Medicine Combined With Thermal and Cold Ablation for Early-stage Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ming Li, senior doctor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021SH10
Record Dates: First submitted 2021-06-29; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Non-small Cell Lung Cancer Stage I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional Chinese medicine combined with thermal or cold ablation (Experimental)
  Interventions: Combination Product: traditional Chinese medicine and ablation in the primary tumor sites
- thermal or cold ablation (Active Comparator)
  Interventions: Procedure: ablation

INTERVENTIONS:
Combination Product: traditional Chinese medicine and ablation in the primary tumor sites — Patients will be treated with traditional Chinese medicine and ablation in the primary tumor sites
  Arms: traditional Chinese medicine combined with thermal or cold ablation
Procedure: ablation — Patients will be treated with ablation in the primary tumor sites
  Arms: thermal or cold ablation

SUMMARY:
Lung cancer is the leading cause of cancer related mortality. At present, surgical treatment is the main choice for early-stage lung cancer. Even after surgery, the 5-year recurrence rate is still as high as 18.4%-24%. Traditional Chinese medicine combined with thermal and cold ablation could be an alternative treatment. Small sample clinical cases verified that this therapy could be an efficacy and safe treatment in a short period. The primary aim of this trial is to evaluate the efficacy of traditional Chinese medicine combined with thermal and cold ablation for patients with stage I non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient can understand and voluntarily join the study, sign the informed consent form, and the compliance is good.
* Patients with lung nodule.
* Maximum diameter of lung nodule ≥8mm.
* The pathology of lung nodules biopsy was non-small cell lung cancer.
* I period according to the eighth edition of the TNM staging period.
* No mediastinal lymph node metastasis.
* Eastern Cooperative Oncology Group performance status of 0 to 1.
* No prior anticancer treatments including surgery, radiation,chemotherapy or local treatments.
* Sufficient organ functions.

Exclusion Criteria:

* Patients with previous use of various hormones, immunosuppression or autoimmune diseases.
* Women during pregnancy or breast-feeding.
* Patients with severe heart, lung, kidney disease or other systemic diseases
* Patients with severe hemorrhagic diseases.
* Patients with a history of drug abuse or mental illness.
* Other conditions that the investigator has determined are not suitable for participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years after ablation
  Response were evaluated in this study using the revised international criteria (1.1) proposed by the RECIST (Response Evaluation Criteria in Solid Tumours) committee. BEST RESPONSE from the start of study treatment until the end of treatment were reported. Objective response rate is the sum of CR + PR divided by the total number of patients in each group.

SECONDARY OUTCOMES:
DFS | 2 years after ablation
  The time interval from the first medication to the observation of recurrence or metastasis, or death from any cause (calculated based on the previous event). Patients who have not relapsed, metastasized or died at the time of the data cutoff, and those who were lost to follow-up in the study will be counted on the date of their last tumor evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China